CLINICAL TRIAL: NCT02271529
Title: Zilver Paclitaxel(PTX) Thumbwheel Delivery System
Brief Title: Zilver PTX Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-14
Record Dates: First submitted 2014-10-17; First posted 2014-10-22 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Peripheral Vascular Disease
Keywords: Peripheral Vascular Disease; Femoral Artery; Drug-Eluting Stent
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug Eluting Stent (Experimental): Zilver® Paclitaxel(PTX)® Drug-Eluting Peripheral Stent
  Interventions: Device: Zilver® PTX® Drug-Eluting Peripheral Stent

INTERVENTIONS:
Device: Zilver® PTX® Drug-Eluting Peripheral Stent — Treatment of symptomatic vascular disease of the native above-the-knee femoropopliteal arteries.

SUMMARY:
The objective of this study is to evaluate the performance of the Zilver PTX stent thumbwheel delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Patient has symptomatic vascular disease of the native above-the-knee femoropopliteal arteries
* Patient has atherosclerotic lesion of the above-the-knee femoropopliteal artery

Exclusion Criteria:

* Patient is < 18 years of age
* Patient unable to complete required follow-up assessments
* Patient unwilling to sign and date the informed consent
* Simultaneous participation in another investigational drug or device study
* Pregnant, breastfeeding or planning to become pregnant in the next 5 years
* Additional medical/anatomical restrictions as specified in the Clinical Investigation Plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MD, Principal Investigator — Auckland District Health Board
Locations (6):
- Australia (2):
  - Frankston Hospital, Frankston
  - Princess Alexandra Hospital, Woolloongabba
- Universitäts-Herzzentrum Freiburg - Bad Krozingen GmbH, Bad Krozingen, Germany
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington

RESULTS

PARTICIPANT FLOW:
Groups:
- Zilver® Paclitaxel(PTX)® Drug-Eluting Peripheral Stent: Treatment of symptomatic vascular disease of the native above-the-knee femoropopliteal arteries.
Period: Overall Study
Arm/Group | Zilver® Paclitaxel(PTX)® Drug-Eluting Peripheral Stent
Started | 40
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zilver® Paclitaxel(PTX)® Drug-Eluting Peripheral Stent
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Stent Length Upon Deployment
Time Frame: Immediately following completion of the stent placement procedure
Population: There were 63 implanted stents, an assessment of stent length change was not available for 2 stents.
Measure: Mean (Standard Deviation); unit: percentage of change in stent length
Units Other Than Participants: Stents
Arm/Group | Zilver® Paclitaxel(PTX)® Drug-Eluting Peripheral Stent
Number analyzed (Participants) | 39
Number analyzed (Stents) | 61
percentage of change in stent length | -1.0 (2.1)
Statistical Analysis 1: Comparison: Zilver® Paclitaxel(PTX)® Drug-Eluting Peripheral Stent; Test type: Non-Inferiority or Equivalence — Under the assumption that the mean percent change in stent length upon deployment being 0.2% with a standard deviation of 4%, type I error of 0.05, and two one-sided t-tests, a sample size of at least 30 stents provides power > 0.90 to determine that the mean length change of stents deployed with the thumbwheel delivery system is within +/-10%; p < 0.01, two one-sided t-tests; Mean percent change = -1.0, 95% CI 2-sided [-1.5 to -0.4]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Zilver® Paclitaxel(PTX)® Drug-Eluting Peripheral Stent
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilver® Paclitaxel(PTX)® Drug-Eluting Peripheral Stent (N=40)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Vascular injury requiring intervention (Vascular disorders) | 1 (1)
Extensive metastatic disease of the abdomen and pelvis (Gastrointestinal disorders) | 1 (1)
Ooze from left groin access site (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days